CLINICAL TRIAL: NCT07407114
Title: Effects of Different Stimuli Applied to the Forearm Flexor Muscles on Muscle Activation, Hand Grip Strength, Reaction Time, and Hand Function
Brief Title: Effects of Different Stimuli on Muscle Activation, Hand Grip Strength, Reaction Time, and Hand Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lokman Hekim University (Other Government)
Responsible Party: Principal Investigator, Seda BAKTIR, Assist. Prof., Lokman Hekim University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: LHU-FTR-ZSBD-06
Record Dates: First submitted 2026-01-29; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Upper Extremity Dysfunction
MeSH Terms: interventions — Ice; Vibration

STUDY DESIGN:
Intervention Model Description: Healthy young participants.
Who Masked: Outcomes Assessor
Masking Description: The assesors are blind to study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group-Ice (Experimental): Cold Application (Ice Therapy):
  Ice application will be administered to the forearm flexor muscle group. The application will be performed using a gel pack available in the Physiotherapy and Rehabilitation Laboratory. The gel pack will be kept in a refrigerator for at least 20 minutes prior to application. The pack will be placed between wet towels and applied continuously to the target area for 3 minutes (reference).
  Interventions: Other: Ice
- Group-Vibr (Active Comparator): Vibration Application:
  Vibration therapy will be applied using the Compex Fixx 1.0 device. The device has three different vibration speed levels. In the present study, vibration will be applied to the forearm flexor muscle groups for 3 minutes at the first speed level (1500 RPMs; Power: W / Voltage: 12.0 V / Current: 0.28 A / Sound level: 57-60 dB).
  Interventions: Other: Vibration
- Croup-Cont (No Intervention): Control Group:
  In the present study, the control group will be planned as a passive control group, and no intervention will be applied. After the baseline measurements, participants will rest in the intervention room for 3 minutes (equal to the duration of the other interventions), followed by post-intervention assessments conducted in the assessment room.

INTERVENTIONS:
Other: Ice — Ice will be used as sensory stimulant in this group.
  Arms: Group-Ice
Other: Vibration — Vibration will be used as sensory stimulant in this group.
  Arms: Group-Vibr

SUMMARY:
The study will include three separate intervention groups: an ice application group, a vibration application group, and a control group. Accordingly, three groups were randomly generated using the Research Randomizer software.

To determine the group allocation of the participants, individuals will be asked to draw a number from a bag containing numbers, each written only once. The intervention corresponding to the drawn number will be applied to the participant.

All interventions will be administered by the researcher Demet Öztürk, while the outcome measurements will be evaluated by the researchers Seda Baktır Doğan and Mustafa Sarı. The interventions and assessment procedures will be conducted in separate rooms in order to ensure assessor blinding.

Participants included in the study will first complete a Demographic Data Form. This form will record demographic information including age, sex, body weight, height, dominant side, alcohol consumption status, medical history, and family history.

Following the relevant tactile stimulus application, participants' hand grip strength, muscle activation, hand function, and upper extremity reaction time will be assessed.

DETAILED DESCRIPTION:
Cold Application (Ice Therapy):

Ice application will be administered to the forearm flexor muscle group. The application will be performed using a gel pack available in the Physiotherapy and Rehabilitation Laboratory. The gel pack will be kept in a refrigerator for at least 20 minutes prior to application. The pack will be placed between wet towels and applied continuously to the target area for 3 minutes (reference).

Vibration Application:

Vibration therapy will be applied using the Compex Fixx 1.0 device. The device has three different vibration speed levels. In the present study, vibration will be applied to the forearm flexor muscle groups for 3 minutes at the first speed level (1500 RPMs; Power: W / Voltage: 12.0 V / Current: 0.28 A / Sound level: 57-60 dB).

Control Group:

The control group will be planned as a passive control group, and no intervention will be applied. After the initial measurements, participants will rest in the intervention room for 3 minutes (equal to the duration of the other interventions), followed by post-intervention assessments conducted in the assessment room.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult individuals aged between 18 and 35 years
* Voluntary participants who have read and signed the informed consent form will be included in the study

Exclusion Criteria:

* Individuals with any systemic, inflammatory, neurological, or degenerative disease affecting the upper extremity
* Individuals with acute inflammation or inflammatory disorders, acute thrombosis, cardiovascular/circulatory diseases, migraine, or epilepsy
* Individuals with a history of trauma or surgery involving the upper extremity within the past year
* Individuals who have started using medications within the last 6 months that may affect the nervous or musculoskeletal systems
* Individuals with implanted metallic foreign bodies in the upper extremity
* Individuals with a pacemaker
* Individuals with circulatory disorders in the upper extremity
* Individuals with any diagnosed sensory impairment
* Individuals with any health condition (e.g., visual or cognitive impairment) that may prevent the proper completion of the assessments

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2023-03-30 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
Muscle Activation Measurement | The evaluations were performed at baseline and immediately post-intervention.
  Surface (non-invasive) electromyography (EMG) will be used to assess muscle activation using the Trigno™ Wireless System (Delsys Inc., USA). EMG recordings will be obtained from the flexor carpi radialis, flexor carpi ulnaris, flexor digitorum superficialis, and flexor digitorum profundus muscles. Electrode placement on the target muscles will be determined according to the SENIAM recommendations and previously published studies.
Hand Grip Strength Measurement | The evaluations were performed at baseline and immediately post-intervention.
  Gross hand grip strength will be assessed using an electronic hand dynamometer (Baseline 12-0286 Electronic Smedley Hand Dynamometer, 200 lbs capacity). Measurements will be performed according to the standard testing protocol recommended by the American Society of Hand Therapists. Participants will be seated upright in a chair with back support, with the shoulder adducted and in a neutral position, the elbow flexed at 90°, and the forearm and wrist in a neutral position. The dynamometer will be held vertically, perpendicular to the floor. Participants will be instructed to hold the dynamometer with one hand and squeeze it as forcefully as possible.

SECONDARY OUTCOMES:
Hand Function Measurement | The evaluations were performed at baseline and immediately post-intervention.
  Hand functional performance will be assessed using the Nine-Hole Peg Test (NHPT), a widely used and valid, reliable dexterity test. The test consists of a square platform with nine holes and nine cylindrical pegs that fit into the holes. During the test, participants will be instructed to place the nine pegs into the holes as quickly as possible and, upon completion, immediately remove them and return them to the container.
Upper Extremity Reaction Time Measurement | The evaluations were performed at baseline and immediately post-intervention.
  Upper extremity reaction time will be assessed using the Nelson Visual Hand Reaction Test. Participants will be seated on a chair with the forearm and hand resting comfortably on a table. The thumb and index finger will be positioned approximately 8-10 cm beyond the edge of the table, with the dorsal surfaces of the thumb and index finger parallel to each other in a ready position.The numerical value corresponding to the upper edge of the thumb at the point where the ruler is caught will be read and recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Lokman Hekim University, Ankara, Cankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No